CLINICAL TRIAL: NCT00554697
Title: Influence of Diabetes Mellitus Type II on Tissue Oxygenation in the Perioperative Period
Brief Title: Diabetes Mellitus Type II and Tissue Oxygenation
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit subjects
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrea Kurz, Principal Investigator, The Cleveland Clinic
Other Study IDs: 07-782
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type II
Keywords: tissue oxygenation; perioperative; outcome
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
The purpose of this study is to determine whether diabetics have decreased amounts of oxygen in the skin compared to non-diabetic individuals, and if the amount of oxygen in the skin changes when given more oxygen to breathe around the time of surgery. To do this, the investigators will be measuring the amount of oxygen in the skin of diabetic and non-diabetic individuals who will be undergoing abdominal surgery lasting 2-4 hours. These measurements will be taken at three different times.

DETAILED DESCRIPTION:
The goal is to test the hypothesis that: 1) perioperative subcutaneous oxygenation (PsqO2) is lower in diabetic than non-diabetic patients; and, 2) supplemental oxygen provides less benefit in diabetic than non-diabetic patients.

We propose a prospective case-control study which will include 30 Type II diabetics matched for age, sex, and race to 30 non-diabetic controls. Patients will be preselected from a population undergoing abdominal surgery and given supplemental inspired oxygen of 30 - 80% to PaO2 of approximately 150mmHg and/or 300mmHg at three timepoints in the perioperative period. PsqO2 will be measured with an IV-sized probe inserted through a small incision made in the skin. Data will be recorded and analyzed using unpaired two tailed t-test, Wilcoxon's ranked sum test, or repeated-measures analysis of variance (ANOVA) test as appropriate.

ELIGIBILITY:
Inclusion criteria:

We will include 30 patients who have more than a five-year history of insulin-dependent type-2 diabetes mellitus and 30 non-diabetic patients meeting the following criteria:

* 35 - 65 yrs old
* BMI < 30
* ASA class I - III
* Abdominal surgery scheduled to last between 2- 4 hours

For Non-diabetic group:

previous BMP within the last year demonstrating glucose < 126mg/dL

For Diabetic group:

* DMII defined as fasting plasma glucose of > 126 mg/dL at time of diagnosis, now requiring insulin
* At least one diabetes associated vasculopathy: coronary artery disease, diabetic nephropathy, hypertension, diabetic retinopathy, diffuse neuropathy, peripheral vascular disease, or a history of stroke

Exclusion Criteria:

* Pregnant
* Immunocompromised: HIV/AIDS, on immunosuppressant therapy for any reason, or post-organ transplantation.
* Infection or fever, or on glucocorticoids
* Malignancy currently requiring radiation or chemotherapy
* Liver or renal failure
* Pancreatic insufficiency, dysautonomia, thyroid disease, Raynaud's syndrome, pathologic Allen-test, or any coagulopathies
* Respiratory disease affecting ability to reach PaO2 of 300mmHg: COPD, emphysema, cystic fibrosis, asthma, pneumonia, PE
* Smoker within the past 6 months or current alcohol abuse
* Allergy to local anesthetic
* For diabetics: DMI, other specific subtype, and gestational diabetics
* We will also exclude patients with epidural catheter, to avoid the influence of regional anesthesia on tissue oxygenation [37, 38].

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include 30 patients who have more than a five-year history of insulin-dependent type-2 diabetes mellitus and 30 non-diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Diabetes Mellitus Type II and Tissue Oxygenation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, M.D., Study Chair — The Cleveland Clinic; Andrea Kurz, M.D., Principal Investigator — The Cleveland Clinic